CLINICAL TRIAL: NCT06631482
Title: Randomized Controlled Trial Comparing HPI and Elevated Threshold Monitor Alarms in Preventing Intraoperative Hypotension
Brief Title: Comparison Bewteen Intraoperative HPI vs. High Mean Arterial Pressure Threshold
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202406137RIND
Record Dates: First submitted 2024-09-18; First posted 2024-10-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Hypotension During Surgery
Keywords: HPI; intraopeartive hypotension; overtreatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HPI Group (Experimental): Use the hypotension predictive index (HPI)-guided protocol to prevent intraoperative hypotension, initiating treatmentusing the fluid administration or intravenous norepinephrine infusion to keep intraoperative HPI below 85.
  Interventions: Device: Maintain HPI < 85
- 73mmHg MAP Alarm Group (Active Comparator): Intraoperative maintenance of the mean arterial pressure (MAP) at 73 mmHg or higher by using the fluid administration or intravenous norepinephrine infusion.
  Interventions: Drug: Maintain MAP>=73

INTERVENTIONS:
Device: Maintain HPI < 85 — Protocolized treatment with fluid administration, norepinephrine, and dobutamine to prevent intraoperative hypotension. The two arms are triggered by different alarms: one from a traditional monitor with an elevated MAP threshold of 73 mmHg, and the other from an HPI threshold of 85.
  Arms: HPI Group
Drug: Maintain MAP>=73 — Protocolized treatment with fluid administration, norepinephrine, and dobutamine to prevent intraoperative hypotension. The two arms are triggered by different alarms: one from a traditional monitor with an elevated MAP threshold of 73 mmHg, and the other from an HPI threshold of 85.
  Arms: 73mmHg MAP Alarm Group

SUMMARY:
Intraoperative hypotension (IOH) is a common and serious complication during surgery, closely associated with poor postoperative outcomes. Traditionally, anesthesiologists rely on real-time physiological parameters and alarms to monitor blood pressure, but the low alarm thresholds may lead to delayed interventions. The Hypotension Prediction Index (HPI) is a novel predictive tool that uses arterial waveform signals and advanced algorithms to forecast hypotensive events in advance. Recent observational studies have shown that HPI's accuracy in predicting hypotension is highly consistent with setting the physiological monitor's alarm threshold to 73 mmHg. This study will compare the effectiveness of HPI and a raised alarm threshold of 73 mmHg in preventing IOH. While HPI is promising with its AI-assisted approach to patient care, its high cost due to the advanced technology raises concerns. If its accuracy is comparable to simply raising the traditional monitor threshold, it may not lead to substantial changes in clinical practice.

DETAILED DESCRIPTION:
Intraoperative hypotension (IOH) is a significant complication that affects surgical patients, potentially leading to adverse outcomes postoperatively. Standard practices involve relying on monitoring devices with low alarm thresholds for blood pressure, which may result in delayed interventions. The Hypotension Prediction Index (HPI) offers a predictive approach by analyzing arterial waveform signals and using complex algorithms to detect potential hypotensive episodes early. Recent observational studies have suggested that HPI's accuracy in predicting hypotension aligns closely with raising the physiological monitor alarm threshold to 73 mmHg. To further investigate this, this study will compare the effects of setting a traditional monitor alarm threshold at 73 mmHg with using HPI to prevent IOH.

In this study, patients will be randomly assigned to two groups. In the HPI group, interventions will be initiated when the HPI value exceeds 85. These interventions will follow a protocol that includes fluid administration, norepinephrine, and dobutamine to prevent hypotension. The control group will have their alarm threshold set at 73 mmHg. For these patients, interventions will be based on stroke volume variation (SVV) and clinical judgment, utilizing fluid and norepinephrine as needed. HPI is an attractive AI-based tool for medical care, but its high cost due to advanced technology raises questions. If its accuracy proves to be similar to simply raising the alarm threshold to 73 mmHg, it may not lead to meaningful changes in clinical practice. The study aims to compare the efficacy of these two methods in reducing the incidence of IOH.

ELIGIBILITY:
Inclusion Criteria:

* A: Patients undergoing surgeries requiring general anesthesia lasting more than two hours, and requiring continuous arterial blood pressure monitoring via arterial catheter according to standard medical practice. This includes:

ASA Class II or higher. Estimated surgery duration of three hours or more. High cardiovascular risk, such as poorly controlled hypertension, diabetes, coronary artery disease, chronic kidney disease, or chronic emphysema.

* B: Patients aged 18 years or older.

Exclusion Criteria:

* ASA Class I: Patients with mild systemic disease.
* Pregnancy: Pregnant women.
* End-stage renal disease: Patients with eGFR below 30 ml/min/1.73 m².
* Cardiac shunt: Presence of intracardiac shunt.
* Severe arrhythmias: Including supraventricular tachycardia (heart rate >100 bpm), ventricular tachycardia, or ventricular fibrillation.
* Factors affecting SVV accuracy: Conditions such as atrial fibrillation (A-Fib) or thoracic surgery that can invalidate stroke volume variation (SVV) measurements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Time-Weighted Average (TWA) for MAP below 65 mmHg During Surgery | From the start of surgery to the end of surgery, approximately up to 12 hours, depending on the duration of the operation.
  The primary outcome will assess the time-weighted average (TWA) for both groups, comparing the duration and magnitude of mean arterial pressure (MAP) below 65 mmHg during surgery. This will help determine the effectiveness of the interventions in preventing intraoperative hypotension and hypertension.
Comparison of Time-Weighted Average (TWA) for MAP above 100 mmHg During Surgery | From the start of surgery to the end of surgery, approximately up to 12 hours, depending on the duration of the operation.
  The primary outcome will assess the time-weighted average (TWA) for both groups, comparing the duration and magnitude of mean arterial pressure (MAP) above 100 mmHg during surgery. This will help determine the effectiveness of the interventions in preventing intraoperative hypotension and hypertension.

SECONDARY OUTCOMES:
30-day mortality rate | From the day of surgery to 30 days postoperatively.
  30-day mortality rate from the day of the surgery.
dosage of intraoperative interventions (such as vasopressors and fluids) | During the surgery (from induction of anesthesia to the end of surgery, approximately up to 12 hours, depending on the duration of the surbery).
  The type, and dosage of intraoperative interventions (such as vasopressors and fluids) administered during surgery.
hospital stay | Approximately 7 days from the date of enrollment
  Total hospital stay duration in days.

CONTACTS AND LOCATIONS:
Overall Officials: Tsung Ta Wu, MD., Principal Investigator — National Taiwan University Hospital Hsinchu branch
Locations (2):
- Taiwan (2):
  - National Taiwan University Hosipital, Taipei
  - National Taiwan University Hospital Hsin-Chu Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulder MP, Harmannij-Markusse M, Fresiello L, Donker DW, Potters JW. Hypotension Prediction Index Is Equally Effective in Predicting Intraoperative Hypotension during Noncardiac Surgery Compared to a Mean Arterial Pressure Threshold: A Prospective Observational Study. Anesthesiology. 2024 Sep 1;141(3):453-462. doi: 10.1097/ALN.0000000000004990. PMID 38558038
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315